CLINICAL TRIAL: NCT00122005
Title: Phase I/II Study of Human GM-CSF Gene-Transduced Irradiated Prostate Allogeneic Cancer Cell Vaccines (GVAX®) in Advanced Prostate Cancer Patients Made Lymphopenic and Infused With Autologous Peripheral Blood Mononuclear Cells
Brief Title: GVAX in Advanced Prostate Cancer Patients Made Lymphopenic
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Providence Health & Services (Other)
Collaborators: Providence Cancer Center, Earle A. Chiles Research Institute (Other); Cell Genesys (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PPMC-EACRI-IRB-02-119; DOD Grant #DAMD17-03-1-0097
Record Dates: First submitted 2005-07-18; First posted 2005-07-21 (Estimated); Last update posted 2009-02-24 (Estimated); Status verified 2009-02

CONDITIONS: Prostate Cancer
Keywords: Metastatic; Prostate; Advanced; Cancer; GVAX; Vaccine
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis; Neoplasms

INTERVENTIONS:
Biological: GM-CSF gene transduced allogeneic vaccine GVAX

SUMMARY:
Androgen (a male sex hormone) deprivation is the standard therapy for metastatic prostate cancer and results in regression or control of disease in 80-85% of patients. This hormone therapy results in a progression-free survival of 12-18 months and overall survival of 24-30 months. However, all patients ultimately develop hormone-refractory prostate cancer (HRPC). Management of HRPC patients is a significant challenge for both patient and physician. Neither past nor current chemotherapy regimens have shown curative potential in patients with HRPC. Thus new treatment strategies are a high priority.

A major focus of new treatment strategies is to enlist the aid of the immune system, particularly the development of prostate cancer vaccines. There has been a number of studies using dendritic cell based vaccines and the treatment has been well tolerated. Specific T-cell immune responses have been observed and occasional evidence for tumor regression. A reduction in serum prostate-specific antigen (PSA) has been observed as well. Lengthening the time-to-progression and delays in the onset of bone pain have been observed in subsets of patients with HRPC.

The initial preclinical observations suggesting that a granulocyte-macrophage colony-stimulating factor (GM-CSF) gene transduced allogeneic (GVAX) prostate cancer vaccine may be efficacious in poorly immunogenic cancers were reported.

The objective of this study is to evaluate the safety and immunologic effects of vaccinations with Allogeneic Prostate GVAX® (CG1940 & CG8711) in patients made lymphopenic by treatment with chemotherapy and infused with autologous peripheral blood mononuclear cells (PBMC). Clinical observations and laboratory measurements will be monitored to evaluate safety, toxicity and immune responses. Additionally, the effects of treatment on serum PSA levels and tumor response will be evaluated.

DETAILED DESCRIPTION:
Other investigators have focused on tumor cell-based vaccine strategies using either allogeneic or autologous tumor cells. Vaccines derived from allogeneic melanoma tumor cell lines are associated with no clinically significant toxicity when given alone.

Most tumor cell line vaccines are lethally irradiated, but not genetically modified. However, a newer generation of tumor vaccines that have been genetically modified to enhance tumor-associated antigen presentation to patient T cells have reached early clinical trials. Based on extensive preclinical studies and clinical allogeneic prostate cancer vaccine data, a strong impression exists that ex vivo GM-CSF gene transfer may make human prostate cancer cell lines more potent in inducing clinically relevant antitumor immune responses in men with micrometastatic prostate cancer.

In the early clinical studies of irradiated GM-CSF-secreting autologous cancer cell vaccine treatment of advanced kidney cancer and advanced melanoma, immune responses elicited by vaccination appeared dependent on both the vaccine cell dose administered and the level of GM-CSF secretion by the vaccine cells. A significant fraction of the nearly 50,000 men each year who suffer from life-threatening prostate cancer will not be candidates for autologous tumor vaccine treatments simply because an insufficient number of autologous prostatic carcinoma cells will be available after surgery. These men may benefit from an allogeneic GM-CSF-gene-transduced prostate cancer vaccine.

Theoretically, autologous prostate cancer cells may be the best source of prostate cancer antigens for eliciting therapeutically useful immune responses. However, evidence has accumulated to suggest that allogeneic prostatic carcinoma cells might also serve as useful sources of prostate cancer antigens for prostate cancer vaccine construction. One theoretical concern about the use of allogeneic prostate cancer cells to prime antigen specific T-cell immunity is whether cytolytic T lymphocytes (CTLs) restricted to the HLA molecules of the patient's tumors can be primed by vaccine cells expressing different (allogeneic) HLA molecules. Recent work has shown that the GM-CSF gene transduced tumor cells do not directly prime MHC class I restricted CTLs but are broken down by the recipient's antigen-presenting cells, which process and present these antigens on their HLA molecules to prime T cells. In fact, tumor cells that do not express any MHC class I molecules are nevertheless capable of generating systemic antitumor immunity that is comparable to their MHC class I positive counterparts.

Phase I and II studies of the allogeneic prostate cancer vaccine have been performed in patients with metastatic prostate cancer. One is a Phase I trial of CG1940 alone and one is a phase I/II trial of CG1940 and CG8711 using the AAV GM-CSF vaccine cells. These trials are currently in progress to evaluate safety and time to progression by PSA and bone scan. In these trials the vaccines are administered at dose levels of 5 x 10^7, 1 x 10^8, 2 x 10^8, or 3 x 10^8 cells every 2 or 4 weeks for 3 to 12 vaccinations and a 5 x 10^8 cell prime vaccination followed by a 3 x 10^8 cell boost vaccination every 2 weeks for a total of 13 vaccinations. Preliminary analysis of the 12 patients enrolled in the phase I trial shows one patient with stable disease. Eighty patients have been enrolled in the phase II trial. Sixty-five of these patients in the phase II trial have been followed for a median of 4 months. One of these patients had a partial PSA response, and 10 maintained stable PSAs. Follow-up bone scans were obtained in 33 patients. One patient showed improvement in metastatic lesions on his bone scan, and 12 patients maintained stable disease on bone scans. ICTP was assayed at Treatment 1, Treatment 4, and at the First Follow-Up Visit in fifteen patients. The ICTP level decreased in five patients (33%) of whom two had undetectable levels after vaccine treatment. This normalization of osteoclast activity suggests a novel mechanism of immunotherapy in metastatic prostate cancer.

As of November 29, 2004, 188 patients have received the prostate GVAX vaccine. In summary, these phase I and II trials showed that CG1940 and CG8711 has an excellent safety profile. As of January 24, 2005, a phase III trial of prostate GVAX is open at more than 40 medical centers in the USA.

ELIGIBILITY:
Inclusion Criteria:

* Histologically diagnosed adenocarcinoma of the prostate
* Progressive disease
* ECOG performance status of 0 or 1
* Adequate bone marrow, renal and hepatic function
* Castrate levels of testosterone
* May have had local radiotherapy as part of their initial treatment or 28 days after palliative radiotherapy or one chemotherapy treatment for metastatic disease

Exclusion Criteria:

* Transitional cell, small cell or squamous cell prostate cancer
* Systemic steroid therapy within 10-days of enrollment
* Documented history of active autoimmune disease such as lupus, sarcoidosis, rheumatoid arthritis, glomerulonephritis or vasculitis
* Clinically significant active infections
* History of other malignancies over past 5-years (except non-melanoma skin cancer or controlled superficial bladder cancer)
* Uncontrolled medical problems (i.e. neurological, cardiovascular) considered high risk for investigational new drug treatment
* Prior treatment with an investigational drug within 30-days of study entry
* Seropositive for HIV, hepatitis B surface antigen or hepatitis C

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2005-07; Study Completion 2005-07 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety of combined CG1940 & CG8711, chemotherapy with cyclophosphamide +/- fludarabine and hematopoietic reconstitution in patients with advanced hormone-refractory prostate cancer (HRPC)
To explore the effects of different chemotherapy regimens on the immune response of CG1940 & CG8711 vaccinated and reconstituted lymphopenic patients with HRPC
To compare the frequency of tumor vaccine-specific, PSMA-specific T cells, and the titer of vaccine-specific antibodies in Cohorts A-C, compare in Cohorts A-C
To evaluate in vitro sensitization (IVS) methods for their capacity to expand tumor vaccine-specific CD4+ and CD8+ T cells from the peripheral blood
To determine whether the degree of lymphopenia inversely correlates with the expansion of tumor-specific CD4 and CD8 T cells
To evaluate the effects of these procedures on serum PSA levels and tumor response

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Fox, PhD, Principal Investigator — Providence Health & Services
Locations (1):
- Providence Portland Medical Center, Portland, Oregon, United States